CLINICAL TRIAL: NCT05113680
Title: Process Evaluation of the Effectiveness of Two Transdiagnostic Interventions on Emotion Regulation : Compassion Focused Program and Emotion Competence Training Program
Brief Title: Process Evaluation of the Effectiveness of Two Transdiagnostic Interventions on Emotion Regulation
Acronym: INTREC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Marine Paucsik, Clinical PhD Student, University Grenoble Alps
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGrenobleAlps
Record Dates: First submitted 2021-09-20; First posted 2021-11-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Emotion Regulation
Keywords: compassion; emotion regulation; emotional competencies; transdiagnostic
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: compassion focused group, emotional competencies group, control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- compassion (Experimental): compassion focused group based on CFT
  Interventions: Behavioral: compassion focused group
- emotional competencies (Active Comparator): emotional competencies group (based on emotional intelligence)
  Interventions: Behavioral: emotional competencies
- control (No Intervention): control group

INTERVENTIONS:
Behavioral: compassion focused group — Based on compassion focused therapy (CFT) principles practices : soothing breathing rythm, compassionate-self, compassion for shame and self-criticism 12 sessions of 2h each
  Arms: compassion
Behavioral: emotional competencies — Emotional competencies group focused on identification, comprehension, expression, regulation, utilization. practices : TCC, cognitive restructuring, and mindfulness 12 sessions of 2h each
  Arms: emotional competencies

SUMMARY:
Emotional regulation (ER) appears today as a fundamental skill for the adaptation of an individual to his environment. Indeed, functional and efficient ER is crucial for mental well-being, but also for physical health, for the maintenance of satisfying social relationships , and for work performance. Many research studies have shown that difficulties with ER are central to the development of many mental disorders. Consequently, this skill can be the target of psychological interventions , the effectiveness of which can be tested as well as the mechanisms underlying that effectiveness. Various "mechanisms of effectiveness" have been advanced in the literature. Of these, this project will specifically test cognitive flexibility and feelings of self-efficacy.

Although a growing number of interventions attempt to target emotional regulation, few are evaluated in subclinical populations and few are protocolized. Similarly, there is little research evaluating the effectiveness processes of these interventions. To date, two types of interventions show particular promise: emotion competence based interventions and compassion focused therapy. This research will therefore be based on the evaluation of two interventions in a randomized controlled trial: Emotion Competence Training Program and Compassion Focused Program that will take place over 12 two-hour sessions in a subclinical and clinical population.

DETAILED DESCRIPTION:
This study is composed:

* a single case study in a subclinical population
* a randomized controlled study in a subclinical population
* a pilot study in a clinical population

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 inclusive
* Person who can understand, speak and read French
* Person who has been orally informed and has given informed consent to participate in the study
* Affiliated with a social security plan

Exclusion Criteria:

* Score greater than or equal to 14 on the DASS21 scale.
* Current participation in another study regarding emotional regulation
* Participation in positive psychology, mindfulness, or stress management groups for less than 3 months
* Change in psychotropic medication (taking, stopping, or changing dosage) within 2 months prior to study participation
* Substance use
* Person with an intellectual disability.
* Person deprived of liberty by judicial decision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Difficulty in Emotion regulation Scale (DERS, Gratz & Roemer, 2004 | 1week
  The DERS-SF is an 18-item self-report multidimensional scale of emotional regulation skills. The DERS examines six difficulties in emotion regulation: (1) unacceptance of negative emotions, (2) difficulty engaging in goal-directed behaviors in the presence of negative emotions, (3) difficulty controlling impulsive behavior in the presence of negative emotions, (4) limited access to emotion regulation strategies perceived as effective, (5) lack of emotional awareness, and (6) lack of understanding of one's emotions, defined as lack of emotional clarity. Items are scored on a five-point Likert scale. Higher scores indicate the presence of difficulties in emotion regulation. Maximum values is 90 and minimum is 18.

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS21, Henry & Crawford, 2005 | 1week
  The DASS-21 is a self-administered questionnaire that measures the severity of depression (e.g., I couldn't seem to feel anything positive), anxiety (e.g., I worried about situations in which I might panic and make a fool of myself), and stress (e.g., I had trouble calming down) during the past week. Each item is scored from 0 (did not apply to me at all in the past week) to 3 (applied to me very often or most of the time in the past week). Higher scores indicate the presence of symptom of depression, anxiety and stress. Maximum values is 84 and minimum is 21.
Well being scale (PWB; Ryff, 1995) | 1week
  The Psychological Well-Being Scale measures six sub-dimensions of well-being: self-acceptance (a positive attitude toward oneself and others), positive relationships with others (warm, trusting and satisfying relationships), autonomy (independence, ability to follow one's own norms, and resist social pressures), environmental mastery (competence in dealing with the demands of life), life purpose (sense of meaning, goals and direction), and self-fulfillment (openness to new experiences, view of oneself as developing and growing). Higher scores indicate the presence of well being. Maximum values is 108 and minimum is 18.
  We used the 18-item version (3 items per dimension) which is parsimonious and retains good psychometric properties (Ryff & Keyes, 1995).
Self-compassion Short Form Scale (SCS-SF; Neff, 2003) | 1week
  SCS-SF is a 12-item instrument with six subscales assessing elements of self-compassion (i.e., self-kindness, self-judgment, common humanity, isolation, mindfulness, and overidentification). Maximum values is 75 and minimum is 12. The higher the score, the higher the level of self-compassion
Profile of Emotional Competence (PEC, Mikolajczak, Brasseur, & Fantini-Hauwel, 2014) | 1week
  The Emotional Competence Scale is a multidimensional self-assessment scale. It assesses the five fundamental emotional competencies (identification, understanding, expression, regulation, and use of emotions) separately for one's own emotions and the emotions of others. This scale is composed of 50 items (Mikolajczak et al., 2014). Maximum values is 250 and minimum is 50.The higher the scores, the higher the level of emotional competence.

OTHER OUTCOMES:
Belief and expectation about therapy (QCA, Coste, Tarquinio, Rouquette, Montel, & Pouchot, 2019) | 1week
  The questionnaire consists of six items (e.g. How much improvement in your symptoms do you think will occur). Four of the items are measured on a nine-point scale ranging from 1 ("not at all" or "none") to 9 ("very"). Two of the items are measured on an 11-point scale ranging from 0% to 100%. The measure score is summed and ranges from 3 to 27. Higher scores indicate participants having higher credibility or expectation for improvement as a result of the treatment. This scale was completed by the participant during the first measurement time, before they started the interventions.
Satisfaction about therapy and therapist (STTS-R, Oei & Green, 2008) | 12week
  This scale is composed of 13 items assessing three sub-dimensions: (1) the patient's level of satisfaction with the therapy (ST, e.g., I am satisfied with the quality of the therapy I received), (2) the patient's level of satisfaction with the therapist (SWT, e.g., the therapist listened to what I was trying to get across), and (3) overall improvement (e.g., how much did this treatment help with the specific problem that led you to the therapy? ). Maximum values is 75 and minimum is 15. Higher scores indicate that participants were satisfied with the intervention and the therapist

CONTACTS AND LOCATIONS:
Locations (1):
- Marine Paucsik, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol (2021-01-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT05113680/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT05113680/SAP_001.pdf
  • Informed Consent Form (2021-01-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT05113680/ICF_002.pdf